CLINICAL TRIAL: NCT05657977
Title: The Effect of Swaddling Method on Stress Level in Newborns Administration to Nasal CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1234
Record Dates: First submitted 2022-09-01; First posted 2022-12-20 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2022-09

CONDITIONS: Nursing Caries; Newborn Illness; Nurse's Role

STUDY DESIGN:
Intervention Model Description: The one-group, pretest, posttest research design.
Who Masked: Investigator
Masking Description: Just one researcher has to blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pretest (No Intervention): Pretest: The newborn connected to nCPAP will be placed in the supine position and slight extension position on the neck of the newborn to ensure airway patency. The first saliva sample will be taken to measure cortisol level in the 30th minute after the first cry from the newborn who is connected to nasal CPAP. Immediately after the saliva sample is taken in pretest group, the stress level determined by using the "neonatal stress scale", vital signs (respiration, heart rate, oxygen saturation), saliva sample collection time will be recorded on the chart.
- Posttest, swaddling (Experimental): Posttest: The swaddling method will be applied to the newborn after the first saliva sample is taken. A second saliva sample will be taken 30 minutes after swaddling to measure cortisol level. Immediately after the saliva sample is taken in posttest group, the stress level determined by using the "neonatal stress scale", vital signs, saliva sample collection time will be recorded on the chart.
  Interventions: Other: nonpharmacologic intervention (swaddling)

INTERVENTIONS:
Other: nonpharmacologic intervention (swaddling) — Swaddling method;The newborn will be placed on a square fabric blanket in the flexion and abduction position and will be loosely swaddled with a blanket.
  Arms: Posttest, swaddling

SUMMARY:
Transient tachypnea of newborn (TTN) causes 42.5%-60% of non-infectious respiratory distress cases in newborns, it is seen in only 1% of all newborns. In the etiology of TTN, it results from the inability to effectively clear the fetal lung fluid immediately after birth. The most known risk factors of TTN are; prematurity, malpresentation, abnormal birth, premature rupture of the membrane, meconium aspiration, fetal distress, multiple pregnancy, male gender, and low Apgar score. TTN; It typically occurs in term and late preterm newborns within the first two hours of life. For the diagnosis of TTN, respiratory rate >60/min in the first 6-12 hours shows signs of groaning and retraction and improve spontaneously within a few days with 40% or less supportive oxygen therapy.

However, in some rare cases, prolongation of symptoms, noninvasive mechanical ventilation support [nasal continuous positive airway pressure (nCPAP), nonsynchronized nasal intermittent mandatory ventilation (NIMV)] and in some cases invasive (intubated) mechanical ventilation may be required.

Reducing pain and stress in mechanically ventilated infants is important for the prevention of complications that may occur in the future-early period and for recover process. While providing standard health care in the Neonatal Intensive Care Unit (NICU), sources of pain and stress should be identified and controlled. It is necessary to minimize the interventions that will cause pain and stress and to ensure that the newborn copes with the pain. In order to relieve pain and stress, various pharmacological (opioid, non-opioid analgesics) and non-pharmacological (breast milk, pacifier, kangaroo care, flexion posture, swaddling etc.) within the framework of family-centered care and individualized developmental care methods should be used. Pain control is a priority in neonatal nursing care, and it is the nurses; responsibility to select and implement a non-pharmacological intervention to reduce the level of pain. A limited number of studies have been found examining the effects of therapeutic touch and mothers voice on pain and comfort level in newborns, as a behavioral intervention, on relieving stress of body positioning in premature newborns who underwent nCPAP. There was no study found that the swaddling method applied during the procedure in patients followed up on nCPAP had an effect on reducing the stress level of newborns.

DETAILED DESCRIPTION:
The aim of the proposed study is to determine the effect of the swaddling method applied to newborns in noninvasive mechanical ventilators on the stress level, by using the neonatal stress scale and salivary cortisol levels.

Type of the research: The research was planned to be conducted in a single group with a pre-test, post-test pattern experimental type.

Research variables Independent variable: Swaddling method. Dependent Variables: The stress felt by the newborn and the salivary cortisol level

The Hypothesis of the Study: H1: Post-intervention (swaddling method) stress and cortisol levels of newborns on CPAP/noninvasive mechanical ventilator are lower than pre-intervention stress and cortisol levels.

Neonatal Stress Scale: The scale consists of 8 sub-dimensions (facial expression, body color, respiration, activity level, comfortability, muscle tone, extremities, posture), and 3-point Likert type. The items in the scale were graded according to the level of stress and grouped into 8 subgroups. In scoring, each subgroup is evaluated between 0-2 points. A minimum of 0 points and a maximum of 16 points are taken from the scale. The baby whose condition is stable and balanced will get a score of 0 from the scale. A high total score from the scale indicates that the baby's stress level is high.

ELIGIBILITY:
Inclusion Criteria:

* Birth week greater than 35 and birth weight greater than 2000 g,
* Need for nasal CPAP/noninvasive mechanical ventilator,
* Legal guardians' consent to participate in the research,
* Diagnosis of neonatal transient tachypnea after delivery.

Exclusion Criteria:

Mother:

* Taking cortisol-containing medication during the antenatal period
* Taking drugs during the antenatal period
* Being chorioamnionitis
* Metabolic disease (adrenal insufficiency, etc.)

Newborn:

* Amniotic fluid stained with meconium
* Intubation
* Apgar score below 6
* Taking analgesic and narcotic drugs for sedation
* Newborn taking cortisol-containing medication
* Inability to obtain a saliva sample or if it is contaminated with blood
* Signs of nasal injury during noninvasive mechanical ventilation
* Congenital defects that will prevent the wrapping method (spina bifida, gastroschisis, etc.)
* Performing resuscitation
* Newborns with cerebral hypoxia-ischemia
* Non-respiratory (congenital pneumonia, respiratory distress syndrome, congenital heart diseases, hypocalcemia, persistent hypoglycemia) causes,
* Development of neonatal sepsis (If sepsis develops in the newborn within the postnatal 48 hours, the baby will be removed from the sample group. Whole blood, biochemistry, hemoculture, and serology tests are performed at the postnatal 24th hour in the routine practice of the unit. The patient will be excluded from the sample after laboratory tests are performed.)
* Hypocalcemia (low calcium level as a result of the blood gas sample taken while opening the vascular access before nCPAP is connected)

Ages: 10 Minutes to 5 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
First inclusion criteria eligible 20 newborn will be add this study. | up to 2 months
  The saliva-specific Enzyme-Linked ImmunoSorbent Assay (ELISA) will be used for the study, for determine research results (pretest, posttest)

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)